CLINICAL TRIAL: NCT02143180
Title: Accuracy of Real-time Tissue Elastography for Evaluating Hepatic Fibrosis in Chronic Hepatitis: a Prospective Multicenter Study.
Brief Title: Accuracy of RTE for Evaluating Hepatic Fibrosis in Chronic Hepatitis: a Prospective Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Rongqin Zheng, professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ThirdSunYatSen
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Hepatitis
Keywords: real-time tissue elastography; hepatic fibrosis
MeSH Terms: conditions — Hepatitis, Chronic; Liver Cirrhosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our study is a prospective multicenter research and the aim is to explore a variety of suitable evaluation indicators and criteria for diagnosis of diffuse liver fibrosis, to get the corresponding diagnosis threshold, with the domestic common pathological S stages as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient has a history of chronic hepatitis on clinical diagnosis; 2. Patient undergoed liver biopsy during study time.

Exclusion Criteria:

* 1. Patient cannot receive examination due to critical condition; 2. Patient refuse the examination.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Liver Fibrosis Index (LFI) | During the examination

CONTACTS AND LOCATIONS:
Overall Officials: Rogqin RQ Zheng, doctor, Principal Investigator — The department of Ultrasound, the third affiliated hospital of Sun Yat-son University
Locations (1):
- The department of Ultrasound, the third affiliated hospital of Sun Yat-son University, Guangzhou, Guangdong, China